CLINICAL TRIAL: NCT04580199
Title: Surgical (Total or Hemithyroidectomy)Versus Non Surgical (Ethanol Ablation ,RF Ablation ,Laser Ablation) Management of Thyroid Nodule
Brief Title: Surgical Versus Non Surgical Management of Thyroid Nodule
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Fahd (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Fahd, principle investigator Mahmoud fahd, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: thyroid nodule
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — Thyroidectomy

STUDY DESIGN:
Intervention Model Description: age above 18 male or female manifested thyroid nodule
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- total thyroidectomy (Active Comparator): excision of thyroid gland
  Interventions: Procedure: thyroidectomy
- hemi thyroidectomy (Active Comparator): excision half of thyroid gland
  Interventions: Procedure: thyroidectomy
- ethanol ingection (Active Comparator): ingection of ethanol into thyroid nodule under guidance of ultrasound
  Interventions: Procedure: thyroidectomy
- monopolar radiofrequency (Active Comparator): using radiofrequency for ablation of thyroid nodule
  Interventions: Procedure: thyroidectomy
- laser photocaugulation (Active Comparator): using laser for ablation of thyroid nodule
  Interventions: Procedure: thyroidectomy

INTERVENTIONS:
Procedure: thyroidectomy — to excise the thyroid gland
  Other Names: ethanol ablation RF ablation laser photocaugulation

SUMMARY:
To compare between surgical (hemi thyroidectomy and total thyroidectomy) and non-surgical (medical, ethanol injection,thermal ablation and laser photo coagulation) management of simple thyroid nodule regarding:

* Outcome of every type of management
* Feasibility of minimally invasive technique in management of simple thyroid nodule in Asyut university
* Complication of every type of management

DETAILED DESCRIPTION:
Thyroid nodules are very common in clinical practice; they are discovered by palpation in 3-7% and by ultrasound (US) in about 50% of the general population. The majority of thyroid nodules are benign and asymptomatic. The main management of benign thyroid nodules is observation and follow-up; however, a minority of them (10-15%) increase in size over time and may induce symptoms or cosmetic issues. Surgical excision has been established as a treatment for symptomatic benign thyroid nodules. thyroidectomy for benign thyroid disease continues to remain controversial, as there are many conflicting data published in the literature regarding the risk of hypothyroidism and recurrent laryngeal nerve injury stratified to indications for surgery, extent of thyroid resection and surgical volume .It carries a 2-10% risk of complications and neck scarring .Thyroid surgery is also costly and may not be appropriate for patients who have a high risk of surgical morbidity.Therefore, image-guided nonsurgical procedures such as ethanol ablation (EA) and thermal ablation have been proposed as alternative and less invasive approaches for the management of benign symptomatic thyroid nodules .These so-called thermoablative methods induce local thermodestruction, leading to nodule shrinkage and improvement of local symptoms. Monopolar radiofrequency ablation (RFA) and EA is widely used as a nonsurgical treatment usually for cystic (i.e., pure cyst) or predominantly cystic benign thyroid nodules (i.e., cystic portion > 50%). There is another method called US-guided percutaneous laser ablation (PLA) is a safe and effective therapeutic option as an alternative to surgery for benign symptomatic nodules

ELIGIBILITY:
Inclusion Criteria:

* complicated thyroid nodule

Exclusion Criteria:

* less than 18 malignant thyroid nodule

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
shrinkage of the thyroid nodule | 2 years
  decrease in the size of thyroid nodule

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin J, Hephzibah J, Cherian AJ, Mathew D, Shanthly N, Oommen R. Is hemi-thyroidectomy adequate in low risk differentiated thyroid cancer? World J Nucl Med. 2019 Apr-Jun;18(2):171-175. doi: 10.4103/wjnm.WJNM_70_18. PMID 31040749
- [Background] Mauri G, Nicosia L, Della Vigna P, Varano GM, Maiettini D, Bonomo G, Giuliano G, Orsi F, Solbiati L, De Fiori E, Papini E, Pacella CM, Sconfienza LM. Percutaneous laser ablation for benign and malignant thyroid diseases. Ultrasonography. 2019 Jan;38(1):25-36. doi: 10.14366/usg.18034. Epub 2018 Sep 17. PMID 30440161
- [Background] Hahn SY, Shin JH, Na DG, Ha EJ, Ahn HS, Lim HK, Lee JH, Park JS, Kim JH, Sung JY, Lee JH, Baek JH, Yoon JH, Sim JS, Lee KH, Baek SM, Jung SL, Kim YK, Choi YJ; Korean Society of Thyroid Radiology (KSThR); Korean Society of Radiology. Ethanol Ablation of the Thyroid Nodules: 2018 Consensus Statement by the Korean Society of Thyroid Radiology. Korean J Radiol. 2019 Apr;20(4):609-620. doi: 10.3348/kjr.2018.0696. PMID 30887743
- [Background] Dobnig H, Amrein K. Monopolar Radiofrequency Ablation of Thyroid Nodules: A Prospective Austrian Single-Center Study. Thyroid. 2018 Apr;28(4):472-480. doi: 10.1089/thy.2017.0547. Epub 2018 Mar 20. PMID 29490593
- [Background] Rahal Junior A, Falsarella PM, Mendes GF, Hidal JT, Andreoni DM, Lucio JFF, Queiroz MRG, Garcia RG. Percutaneous laser ablation of benign thyroid nodules: a one year follow-up study. Einstein (Sao Paulo). 2018 Nov 29;16(4):eAO4279. doi: 10.31744/einstein_journal/2018AO4279. PMID 30517361